CLINICAL TRIAL: NCT01264133
Title: An Open Study to Evaluate the Efficacy, Safety and Sustained Effect of Clevudine Monotherapy or Adefovir and Clevudine Combination in Proportion to Roadmap Concept in Patients With Chronic Hepatitis B
Brief Title: A Study With Clevudine Monotherapy or Adefovir and Clevudine Combination in Patients With Chronic Hepatitis B
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Responsible Party: Byungchul Yoo, Samsung Medical Center
Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CLV-411; CLV-411
Record Dates: First submitted 2010-12-19; First posted 2010-12-21 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — clevudine; adefovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Clevudine, Adefovir — Clevudine 30mg qd or Clevudine 30mg + Adefovir 10mg qd

SUMMARY:
An open study to Evaluate the Efficacy, Safety and Sustained effect of Clevudine monotherapy or Adefovir and Clevudine combination in proportion to Roadmap concept in Patients with chronic hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18 years and older.
2. Patient is documented to be HBsAg positive for > 6 months.
3. Patient is HBV DNA positive with DNA levels ≥ 2,000 IU/mL within 30 days of baseline.
4. Patient has ALT levels >=80 IU/L
5. Patient with compensated liver disease (Patient with chronic B Hepatitis or liver cirrhosis <= 6)
6. Patient who is able to give written informed consent prior to study start and to comply with the study requirements.

Exclusion Criteria:

1. Patient is currently receiving antiviral, immunomodulatory, cytotoxic or corticosteroid therapy.
2. Patients previously treated with interferon, peg-interferon or other immunomodulatory within the previous 6 months.
3. Patients previously treated with clevudine, lamivudine, adefovir, entecavir, telbivudine or any other investigational nucleoside for HBV infection.
4. Patient is coinfected with HCV, HDV or HIV.
5. Patient has a history of ascites, variceal hemorrhage or hepatic encephalopathy.
6. Patient with clinical evidence of decompensated liver disease or hepatocellular carcinoma
7. Patient with previous liver transplantation
8. Patient is pregnant or breast-feeding.
9. Patient has a clinically relevant history of abuse of alcohol or drugs.
10. Patient has a significant immunocompromised, gastrointestinal, renal, hematological, psychiatric, bronchopulmonary, biliary diseases excluding asymptomatic GB stone, neurological, cardiac, oncologic(except HCC)or allergic disease or medical illness that in the investigator's opinion might interfere with therapy.
11. Patient has creatinine clearance less than 60mL/min as estimated by the following formula: (140-age in years) (body weight [kg])/(72) (serum creatinine [mg/dL]) [Note: multiply estimates by 0.85 for women]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-09; Primary Completion 2013-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with HBV DNA levels < 60 IU/mL | 48 week

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea